CLINICAL TRIAL: NCT06857019
Title: Evaluating the Clinical Effectiveness of "Endotracheal Tube Position Anomaly Alerting System"
Acronym: ETPAAS-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20240327
Record Dates: First submitted 2025-02-16; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Critical Care Medicine; Mechanical Ventilation; Radiographic Image Interpretation, Computer-Assisted; Alarms
Keywords: Chest X-ray; Chest radiograph; Endotracheal tube; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ETPAAS (Experimental): Participants receive standard of care, with "Endotracheal Tube Position Anomaly Alerting System" (ETPAAS), in the intensive care unit.
  Interventions: Other: "Endotracheal Tube Position Anomaly Alerting System"
- Control (No Intervention): Participants receive standard of care, without ETPAAS, in the intensive care unit.

INTERVENTIONS:
Other: "Endotracheal Tube Position Anomaly Alerting System" — The "Endotracheal Tube Position Anomaly Alerting System" (ETPAAS) is designed to assist healthcare providers in managing patients receiving mechanical ventilation via an endotracheal tube. This system integrates an artificial intelligence (AI) algorithm that automatically evaluates the appropriateness of endotracheal tube positioning whenever a patient's chest X-ray is uploaded. If the system detects that the distance between the endotracheal tube tip and the carina falls outside the optimal range, it promptly alerts healthcare providers, enabling timely intervention to correct the tube position and enhance patient safety.
  Other Names: ETPAAS
  Arms: ETPAAS

SUMMARY:
The goal of this clinical trial is to determine whether the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) effectively reduces the duration of endotracheal tube malposition in patients admitted to the intensive care unit (ICU). Additionally, the study will assess the clinical impact, usability, and user satisfaction of ETPAAS.

The main questions it aims to answer are:

* Does ETPAAS reduce the duration of endotracheal tube malposition?
* What are healthcare workers' perspectives on the usability and satisfaction of ETPAAS?

Participants will receive standard care, with or without ETPAAS, in the intensive care unit.

Researchers will evaluate the duration of endotracheal tube malposition. Healthcare workers will complete a questionnaire assessing the usability and satisfaction of ETPAAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit
* At least 18 years old

Exclusion Criteria:

* Patients disagree to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of endotracheal tube malposition | from the initial detection of endotracheal tube malposition to its correction, an estimated average of 48 hours

SECONDARY OUTCOMES:
Usability and user satisfaction survey with a questionnaire | through study completion, up to 6 months
Prevalence of endotracheal tube malposition | through study completion, up to 6 months
  Prevalence of endotracheal tube malposition on the first chest radiograph on ICU admission and on the second chest radiograph taken in the ICU
ICU length of stay | from ICU admission to ICU discharge, an estimated average of 7 days
Duration of mechanical ventilation | from intubation to the discontinuation of mechanical ventilation, an estimated average of 5 days
Weaning rate of mechanical ventilation | from intubation to the successful discontinuation of mechanical ventilation, assessed up to 5 months
Accuracy of the ETPAAS | through study completion, up to 6 months
  The accuracy of the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) will be evaluated by comparing its automated assessments of endotracheal tube (ETT) positioning with expert clinical interpretations. Accuracy will be determined based on the system's sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) in detecting ETT malposition. The reference standard will be assessments made by experienced intensivists.
Precision of the ETPAAS | through study completion, up to 6 months
  The precision of the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) will be evaluated by assessing the consistency and reliability of its automated endotracheal tube (ETT) position anomaly detection. Precision will be measured as the proportion of correctly identified malpositioned ETT cases among all positive alerts generated by the system (i.e., positive predictive value, PPV).
Recall of the ETPAAS | through study completion, up to 6 months
  The recall of the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) will be assessed by evaluating its ability to correctly identify cases of endotracheal tube (ETT) malposition. Recall will be quantified as the proportion of true positive cases detected by ETPAAS among all actual cases of ETT malposition, also known as sensitivity. A higher recall value indicates the system's effectiveness in minimizing missed detections and ensuring timely alerts for clinical intervention.
F1 score of the ETPAAS | through study completion, up to 6 months
  The F1 score of the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) will be used to assess the balance between precision and recall in detecting endotracheal tube (ETT) malposition. The F1 score is the harmonic mean of precision and recall. A higher F1 score indicates that ETPAAS effectively identifies ETT malposition with both high accuracy and low false-negative and false-positive rates. This metric provides a comprehensive evaluation of the system's performance in a clinical setting.
Area under the curve (AUC) of receiver operating characteristic (ROC) curve of the ETPAAS | through study completion, up to 6 months
  The Area Under the Curve (AUC) of the Receiver Operating Characteristic (ROC) curve will be used to evaluate the overall diagnostic performance of the Endotracheal Tube Position Anomaly Alerting System (ETPAAS) in detecting endotracheal tube (ETT) malposition. The ROC curve plots the true positive rate (sensitivity) against the false positive rate (1 - specificity) at various classification thresholds. The AUC value ranges from 0 to 1, where:
  * AUC = 1.0 indicates perfect classification performance.
  * AUC = 0.5 suggests no better performance than random chance.
  * Higher AUC values indicate superior discriminatory ability of ETPAAS in correctly distinguishing between correctly positioned and malpositioned ETT cases.
  This metric provides a robust measure of the system's reliability and effectiveness in clinical decision support.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ju Tsai, M.D., Ph.D., Study Director — Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be made available to qualified researchers with academic interests in related fields. All shared data will be coded and stripped of any protected health information. Data sharing will be contingent upon the approval of the request and the execution of all applicable agreements (e.g., a material transfer agreement) before access is granted to the requesting party.
Time Frame: Data requests may be submitted beginning 12 months after the publication of the study article. The data will be accessible for up to 24 months, with extensions considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers conducting independent scientific research. Data access will be granted following the review and approval of a research proposal and a Statistical Analysis Plan (SAP), as well as the execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the Study Director.